CLINICAL TRIAL: NCT02059681
Title: Phase I Trial of Endocavitary Injection of Bone Marrow Derived CD133+ Cells in Ischemic Refractory Cardiomyopathy (RECARDIO Trial)
Acronym: RECARDIO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: A.O.U. Città della Salute e della Scienza (Other); Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Giulio Pompilio, MD PhD, Centro Cardiologico Monzino
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S225/612
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Chronic Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous bone marrow derived-CD133+ cells (Experimental): CD133+ cells (1-12x10^6) suspended in 10 ml physiological saline supplemented with 5% human albumin solution will be injected into the myocardium via the endocardial route; the whole 10 ml solution will be divided into 15-20 injections.
  Interventions: Other: Autologous bone marrow derived-CD133+ cells

INTERVENTIONS:
Other: Autologous bone marrow derived-CD133+ cells — Cell therapy

SUMMARY:
The purpose of this study is to evaluate whether endocavitary intramyocardial injection of autologous bone-marrow-derived CD133+ cells is safe on the basis of number of adverse events, with follow-up assessments extending up to 1 year after enrolment.

DETAILED DESCRIPTION:
This will be a Phase I study investigating the safety and preliminary efficacy of endocavitary injection of bone-marrow-derived CD133+ cells in 15 patients with ischemic heart failure (IHF) not eligible for conventional revascularization. Patients eligible will undergo bone-marrow aspiration. On the day following bone-marrow aspiration patients will undergo fluoroscopy-based endocavitary intramyocardial injections of the target areas previously identified by gated-SPECT/CMR. CD133+ cells suspended in physiological saline supplemented with 5% human albumin solution will be injected into the myocardium via the endocardial route.

After discharge, efficacy follow-up will last 6-months safety follow-up (FU) will be extended up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic heart failure not amenable to any type of revascularization procedure (percutaneous or surgical) as determined by one interventional cardiologist and one cardiovascular surgeon,
2. Canadian Cardiovascular Society Angina functional class III to IV angina and/or symptoms of heart failure (NYHA score IIb to IV) under state-of-the-art maximal medical therapy,
3. Left Ventricular Ejection Fraction between 20% and 45%,
4. Peak V02 ≤ 21 mL/Kg/min,
5. Presence of a reversible perfusion defect ≥ 10% of the left ventricular myocardium (at least 2 segments over 20) as determined by gated-SPECT, 6.18 years ≤ Age ≤ 75 years,

7.Hemodynamic stability, 8.Ability to accomplish a cardiopulmonary exercise testing, 9.Are not pregnant and do not plan to become pregnant during the study. Females with childbearing potential must provide a negative pregnancy test within 1-7 days before intervention and must be using oral or injectable contraception (non-childbearing potential is defined as post-menopausal for at least 1 year or surgical sterilization or hysterectomy at least 3 months before study start), 10.A signed consent form that has been approved by the institutional review board.

Exclusion Criteria:

1. A high-risk acute coronary syndrome (ACS) or a myocardial infarction in the past 3 months,
2. Presence of a documented unstable angina,
3. Left ventricular thrombus, as documented by echocardiography,
4. Evidence of a life-threatening arrhythmia,
5. Presence of any severe mitral valve disease requiring valve replacement or reconstruction,
6. Presence of a mechanical aortic valve,
7. Presence of stenosis of the aortic valve, graded as ≥+2 equivalent to an orifice area of 1,5 cm2 or less,
8. Presence of moderate to severe insufficiency of the aortic valve,
9. A left ventricular wall thickness of <8 mm at the target site for cell injection, as assessed by 2-D echocardiography and/or cardiac MRI,
10. Have a known, serious radiographic contrast allergy,
11. Contraindications to bone-marrow aspiration,
12. Be an organ transplant recipient,
13. Have liver dysfunction, as evidenced by enzymes (AST,ALT) >3x the upper limits of normals,
14. Severe renal failure (creatinine plasma levels > 2.5 mg/dl),
15. A bleeding diathesis (defined as an INR greater than 1,5 not because of a reversible cause, i.e. warfarin),
16. Have an hematologic abnormality without other explanation,
17. Apparent infection (c-reactive protein (CPR)>30 mg/L, fever > 37 °C),
18. An infectious-disease test result positive for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C, treponema pallidum (VDRL), HTLV 1 and 2,
19. Previous or current documented history of leukemia, myeloproliferative or myeloplastic disorders,
20. Have a cardiac condition that limits lifespan to <1 y,
21. A history of malignancy in the past 5 years,
22. Have a history of drug or alcoholic abuse within the past 24 months,
23. Be on chronic therapy with immunosuppressants,
24. Pregnant or lactating status,
25. Any condition that, in the judgment of the investigator, would place the patient at undue risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Safety | 1 year
  The primary objective of this study will be to evaluate whether endocavitary intramyocardial injection of autologous bone-marrow-derived CD133+ cells is safe on the basis of number of adverse events, with follow-up assessments extending up to 1 year after enrolment.

SECONDARY OUTCOMES:
Efficacy | 6 months
  To determine the effects of autologous CD133+ cells as assessed before and 6-months after injection on a) regional myocardial perfusion on the basis of stress gated-SPECT and CMR when available; b) functional capacity on the basis of peak VO2 consumption at CPET.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Pompilio, MD PhD, Principal Investigator — Centro Cardiologico Monzino, IRCCS
Locations (3):
- Italy (3):
  - Azienda Ospedaliera San Gerardo di Monza, Monza, MB
  - Centro Cardiologico Monzino, IRCCS, Milan, MI
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino, TO

REFERENCES:
- [Derived] Bassetti B, Carbucicchio C, Catto V, Gambini E, Rurali E, Bestetti A, Gaipa G, Belotti D, Celeste F, Parma M, Righetti S, Biava L, Arosio M, Bonomi A, Agostoni P, Scacciatella P, Achilli F, Pompilio G. Linking cell function with perfusion: insights from the transcatheter delivery of bone marrow-derived CD133+ cells in ischemic refractory cardiomyopathy trial (RECARDIO). Stem Cell Res Ther. 2018 Sep 14;9(1):235. doi: 10.1186/s13287-018-0969-z. PMID 30217223